CLINICAL TRIAL: NCT06230796
Title: Effects of FES-cycling in Patients With Hemiparesis After Stroke
Brief Title: Effects of Functional Electrical Stimulation Assisted Cycling in Patients With Hemiparesis After Stroke
Acronym: AVCyclES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UGECAM Rhône-Alpes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-01-VR; 2023-A00627-38 (Other: ID-RCB)
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hemiparesis;Poststroke/CVA
Keywords: cycling; exercises; functional electrical stimulation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: In a monocentric, single-blind, randomized, controlled trial, hemiparetic post stroke patients will be randomized to receive FES-induced cycling training or placebo FES cycling.
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FES-cycling (Experimental): 30 minutes of active leg cycling with FES applied to the paretic rectus femoris of quadriceps and to the biceps femoris and semitendinosus muscles and gluteus maximus, 3 times/weeks for 8 weeks
  Interventions: Device: FES-cycling
- SHAM-cycling (Sham Comparator): 30 minutes of active leg cycling with Sham FES applied to the paretic rectus femoris of quadriceps and to the biceps femoris and semitendinosus muscles and gluteus maximus, 3 times/weeks for 8 weeks
  Interventions: Device: SHAM-cycling

INTERVENTIONS:
Device: FES-cycling — 30 minutes of active leg cycling with or without FES applied to the paretic rectus femoris of quadriceps and to the biceps femoris and semitendinosus muscles and gluteus maximus, 3 times/weeks for 8 weeks. During training, participants will be seated on a FES-Cycle (Hepha Bike, Kurage): a cyclo-ergometer (Technogym) combined with a 8 channel controlled stimulator (Motimove-8).
  Arms: FES-cycling
Device: SHAM-cycling — 30 minutes of active leg cycling with SHAM FES applied to the paretic rectus femoris of quadriceps and to the biceps femoris and semitendinosus muscles and gluteus maximus, 3 times/weeks for 8 weeks. During training, participants will be seated on a FES-Cycle (Hepha Bike, Kurage): a cyclo-ergometer (Technogym) combined with a 8 channel controlled stimulator (Motimove-8).
  Arms: SHAM-cycling

SUMMARY:
To determine whether active cycling assisted by functional electrical stimulation (FES) Is more effective than active cycling on cardiovascular fitness in post stroke hemiparesis

DETAILED DESCRIPTION:
Design: In a monocentric, single-blind, randomized, controlled trial, hemiparetic post stroke patients will be randomized to receive FES-induced cycling training or placebo FES cycling.

Setting: Neurologic Rehabilitation Unit Interventions: 30 minutes of active leg cycling with or without FES applied to the paretic rectus femoris of quadriceps and to the biceps femoris and semitendinosus muscles and gluteus maximus, 3 times/weeks for 8 weeks. During training, participants will be seated on a FES-Cycle (Hepha Bike, Kurage): a cyclo-ergometer (Technogym) combined with a 8 channel controlled stimulator (Motimove-8).

In addition to the assigned group treatment, subjects will perform their own standard rehabilitation program.

Participants will be evaluated before training, after training, and at 3 month follow-up visit

ELIGIBILITY:
Inclusion Criteria:

* Adults with Hemiparesis after an unilateral first ever stroke
* Able to walk in security
* Time since stroke within 3 months to 1 year
* Sufficient cognitive function to understand and perform corresponding tasks

Exclusion Criteria:

* Any history of neurological disorders or cardiovascular instability
* High spasticity on ankle, knee, hip muscles
* Inability to exercise on a cyclo-ergometer
* Pacemaker and other contraindications of the use of electrical stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
VO2 peak at 2 months (L/min) | From enrollment to the end of treatment at 8 weeks
  Comparison of the maximum oxygen consumption (VO2 peak in L/min) measured during an incremental maximum stress test on cyclo-ergometer between the end of training (M2) and inclusion (M0).

SECONDARY OUTCOMES:
Maximum power | 2 months
  Comparison of the maximum power (in Watts) developed during the stress test on a cycloergometer between the end of the training (M2) and the inclusion (M0)
Walking ability | 4 months
  walking speed (10m walking test) and distance (6-minute walking test) measured at inclusion, after training (M2) ans follow-up (M4)
quadriceps muscular thickness | 2 months
  quadriceps muscular thickness measured with ultrasound at inclusion aand after the training
Middle Cerebral Artery Blood Flow Velocity During Exercise | 2 months
  Middle Cerebral Artery Blood Flow Velocity During Exercise measured with transcranial Doppler ultrasound at inclusion (M0) and after the training (M2)
Cognitive function | 2 months
  Paper test: Stroop and trail making test at inclusion and after training

CONTACTS AND LOCATIONS:
Locations (1):
- SMR Val Rosay, Saint-Didier-au-Mont-d'Or, France, France